CLINICAL TRIAL: NCT00620334
Title: Predicting the Diagnosis of Asthma Based on History
Brief Title: Predicting the Diagnosis of Asthma
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: RICHARD F LOCKEY, MD, USF
Other Study IDs: COLES
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2008-07

CONDITIONS: Asthma
Keywords: ASTHMA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: ASTHMA:
  PREVOUSLY DIAGNOSED MILD ASTHMA PATIENTS
- 2: CONTROL:
  PATIENTS WHO HAVE NEVER BEEN DIAGNOSED WITH ASTHMA

SUMMARY:
Despite the development of effective medications for treatment, asthma remains a significant contributor of morbidity, mortality, and financial hardship to patients with the disease. An estimated 300 million people worldwide have asthma, making it one of the most common chronic diseases in the world. Asthma accounts for 250,000 deaths per year worldwide, and 1.7 million emergency room visits per year in the United States. Cost of asthma in the United States was an estimated $12.7 billion dollars per year in 1998, and the prevalence is increasing. In 2002, there were 13.9 million outpatient asthma visits to private physician offices and hospital outpatient departments, and 484,000 asthma hospitalizations. Children 5-17 years of age missed 14.7 million school days, and adults missed 11.8 million work days due to asthma in 2002.

There is no single diagnostic test or symptom that defines asthma. Asthma is a syndrome consisting of a constellation of symptoms that include wheeze, cough, shortness of breath, and chest tightness. The diagnosis of asthma takes into account history, physical examination findings, and objective measures of pulmonary function and markers of inflammation. In many cases the diagnosis is not in question, allowing for early recognition and appropriate treatment. In other cases, confounding factors makes the diagnosis both challenging and time consuming for the physician and the patient. According to the National Asthma Education and Prevention Program Expert Panel Report 2, asthma is defined as:

"a chronic inflammatory disorder of the airways in which many cells and cellular elements play a role, in particular, mast cells, eosinophils, T lymphocytes, macrophages, neutrophils, and epithelial cells. In susceptible individuals, this inflammation causes recurrent episodes of wheezing, breathlessness, chest tightness, and coughing, particularly at night or in the early morning. These episodes are usually associated with widespread but variable airflow obstruction that is often reversible either spontaneously or with treatment. The inflammation also causes an associated increase in the existing bronchial hyperresponsiveness to a variety of stimuli."

Airway obstruction and reversibility is measured by pulmonary function testing before and after inhalation of a short acting beta agonist. Airway hyperresponsiveness is measured by methacholine challenge.

Estimates of asthma prevalence are generated by the use of written questionnaires in epidemiologic studies. , One of the difficulties with reliance on questionnaires is that patients often misinterpret the questions or fail to answer the question altogether. In this study, a physician will review the questionnaire with the patient in order to clarify each question.

The goal in this study is to evaluate a simplified set of questions that can be easily implemented into clinical practice that will predict the presence or absence of asthma.

Hypothesis

A simplified questionnaire will predict asthma in adults.

Study Objectives

§ Primary Objective

o To evaluate the predictive value of a questionnaire designed to diagnose asthma in adults

ELIGIBILITY:
Inclusion Criteria:

18-64 years of age at enrollment

* Literacy: The subject must be able to read, comprehend, and record information in English.
* Consent: The subject must have the ability to give informed consent.
* Type of subject: The subject must be seen in the outpatient setting.

Exclusion Criteria:

* Respiratory Instability: Hospitalization for respiratory disease within the last 6 months during study period and prior to Visit 0.
* Respiratory Disease: Current diagnosis of cystic fibrosis, pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, chronic bronchitis, or any other lower respiratory abnormalities other than asthma.
* Prior Treatment of Asthma: Treatment for asthma with any medication (except for short acting inhaled bronchodilators) for 12 months or more prior to Visit 0
* Drug Allergy: Any immediate or delayed hypersensitivity reaction to any beta2-agonist or sympathomimetic drug
* Respiratory Tract Infections: Confirmed or suspected infection of the sinus, middle ear, oropharynx, upper respiratory tract, or lower respiratory tract within 28 days prior to testing
* Other Concurrent Conditions/Diseases: Any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbates during the study. The list of conditions/diseases that will result in exclusion if determined to be clinically significant includes, but is not limited to: cardiac arrhythmia, congestive heart failure, coronary artery disease, Addison's disease, diabetes mellitus, dyspnea by any cause other than asthma, uncontrolled hypertension, hematological, hepatic, neurological, thyroid, peptic ulcer, or renal disease, immunologic compromise, current malignancy, current or quiescent tuberculosis.
* Concomitant Medications:

  1. Beta blockers
  2. Systemic corticosteroids
  3. Angiotensin Converting Enzyme (ACE) inhibitors (Note: Immunotherapy for the treatment of allergies is allowed, provided that the subject has received a constant dose for 30 days prior to Visit 0, and that the same dose will continue throughout the study.)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male or female Females are eligible to participate only if they are currently non-pregnant and non-lactating. All premenopausal women will undergo a urine pregnancy test at the beginning of the study. Female subjects should not be enrolled if they plan to become pregnant during the time of the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the predictive value of a questionnaire designed to diagnose asthma in adults. | UP TO 2 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: RICHARD F LOCKEY, MD, Principal Investigator — University of South Florida
Locations (1):
- USF, Tampa, Florida, United States